CLINICAL TRIAL: NCT04475042
Title: Stratified Treatment to Ameliorate Diastolic Left Ventricular Stiffness in Heart Failure With Preserved Ejection Fraction. A 35-week, Single-center, Prospective, Double-blind, Controlled, Randomized, 2x2 Crossover, Interventional Phase II Study, Investigating the Effect of Treatment With Dapagliflozin 10mg od on Left Ventricular Distensibility in Patients With Early HFpEF.
Brief Title: Stratified Treatment to Ameliorate Diastolic Left Ventricular Stiffness in Heart Failure With Preserved Ejection Fraction
Acronym: STADIA-HFpEF
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mariëlle Scheffer (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Mariëlle Scheffer, Principal Investigator, Onze Lieve Vrouwe Gasthuis
Organization: Onze Lieve Vrouwe Gasthuis (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19.185
Record Dates: First submitted 2020-07-08; First posted 2020-07-17 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Heart Failure, Diastolic
MeSH Terms: conditions — Heart Failure, Diastolic | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Dapagliflozin - washout period - placebo
  Interventions: Drug: Dapagliflozin; Drug: Placebo
- Group B (Active Comparator): Placebo - washout period - Dapagliflozin
  Interventions: Drug: Dapagliflozin; Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin — 10mg od
Drug: Placebo — Placebo

SUMMARY:
A 35-week, single-center, prospective, double-blind, controlled, randomized, 2x2 crossover, interventional Phase II study, investigating the effect of treatment with dapagliflozin 10mg od on Left Ventricular distensibility in patients with early HFpEF.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at time of screening
2. Symptomatic chronic heart failure patients with diagnosis of heart failure and:

   * NYHA class II-IV
   * Preserved systolic Left Ventricular (LV) function, defined by: LV Ejection Fraction (LVEF) ≥ 50% and LV end-diastolic volume index <97 ml/m2
   * Evidence of diastolic LV dysfunction and at least 1 out of the 5 following additional criteria:

     1. H2FPEF score ≥ 6;
     2. HFA-PEFF score ≥ 5;
     3. Pulmonary capillary wedge pressure > 15 mmHg at rest or > 25 mmHg with exercise assessed with right heart catheterization;
3. Cardiac MRI T1 derived extracellular volume <29% at screening
4. Oral diuretics, if prescribed to the patient according to local guidelines and at the discretion of the investigator, should be stable for at least 1 week prior to baseline visit
5. Signed and dated written informed consent in accordance with GCP and local legislation prior to admission to the trial

Exclusion Criteria:

1. Reduced systolic LV function (LVEF < 50%), measured at any time point in the history of the patient
2. Obstructive coronary artery disease with evidence of ischemia
3. Myocardial infarction, coronary artery bypass graft surgery or other major cardiovascular surgery, stroke or TIA in past 90 days prior to screening visit
4. More than mild valve stenosis
5. More than moderate aortic and/or mitral valve regurgitation
6. Cardiomyopathy based on infiltrative diseases (e.g. amyloidosis), accumulation diseases (e.g. hemochromatosis, Fabry disease), muscular dystrophies, cardiomyopathy with reversible causes (stress cardiomyopathy), hypertrophic (obstructive) cardiomyopathy or known pericardial constriction
7. History of mitral valve repair or replacement
8. Atrial fibrillation or atrial flutter with a resting heart rate > 110 bpm at screening
9. Acute decompensation that requires intravenous loop diuretics
10. Systolic blood pressure ≥ 180 mmHg. If SBP > 150 mmHg and < 180 mmHg, the patient should be receiving at least 3 antihypertensive drugs at screening or baseline visit
11. Symptomatic hypotension and/or a SBP < 100 mmHg at screening or baseline visit
12. Impaired renal function, defined as eGFR < 30 ml/min/1.73 m2
13. Indication of liver disease, defined by serum levels of either ALT (SGPT), AST (SGOT), or alkaline phosphatase above 3x upper limit of normal or history of cirrhosis with evidence of portal hypertension
14. Hemoglobin < 9 g/dl at screening
15. Chronic obstructive pulmonary disease, more than GOLD class 2
16. Pulmonary function test with FEV1/FVC < 80%
17. Primary pulmonary arterial hypertension
18. Type 1 Diabetes Mellitus
19. History of ketoacidosis
20. Any documented active or suspected malignancy or history of malignancy within 2 years prior to screening, except appropriately treated basal cell carcinoma of the skin or in situ carcinoma of uterine cervix or low risk prostate cancer (biopsy Gleason score of ≤ 6 and clinical stage T1c or T2a)
21. Current use or prior use of a SGLT-2 inhibitor or combined SGLT-1 and 2 inhibitor within 3 months prior to screening visit. Discontinuation of a SGLT-2 inhibitor or combined SGLT-1 and 2 inhibitor for the purposes of study enrolment is not permitted
22. Pregnancy or lactation
23. Any (clinical) condition that, in the investigator's opinion, would jeopardize patients safety while participating in this trial, or may prevent the patient from adhering to the trial protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Left Ventricular (LV) e' | 13 weeks
  echocardiographically measured
E/e'/LV end-diastolic volume index | 13 weeks
  echocardiographically measured

SECONDARY OUTCOMES:
Kansas City Cardiomyopathy Questionnaire | 13 weeks
6-minute walk test | 13 weeks
Left atrial volume | 13 weeks
  Echocardiographically derived volume
Diastolic parameters | 13 weeks
  Echocardiographically derived function, filling and compliance of Left Ventricular
Left atrial function | 13 weeks
  Echocardiographically derived strain analysis, resevoir, conduit and booster pump function

CONTACTS AND LOCATIONS:
Locations (1):
- OLVG, Amsterdam, North Holland, Netherlands